CLINICAL TRIAL: NCT03887949
Title: Comparison of Three Modes of Ventilation During Robot-assisted Hysterectomy in Trendelenburg Position: Volume Controlled Ventilation, Pressure Controlled Ventilation, and Pressure Controlled Ventilation With Volume Guarantee.
Brief Title: Comparison of Three Modes of Ventilation During Robot-assisted Hysterectomy in Trendelenburg Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Eun Young Park, Associate professor, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-I013
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VCV (Active Comparator): Volume controlled ventilation
  Interventions: Device: Group VCV
- PCV (Active Comparator): Pressure controlled ventilation
  Interventions: Device: Group PCV
- PCV-VG (Experimental): Pressure controlled ventilation with volume guarantee
  Interventions: Device: Group PCV-VG

INTERVENTIONS:
Device: Group VCV — Volume controlled ventilation
  Arms: VCV
Device: Group PCV — Pressure controlled ventilation
  Arms: PCV
Device: Group PCV-VG — Pressure controlled ventilation with volume guarantee
  Arms: PCV-VG

SUMMARY:
Robot-assisted hysterectomy is associated with pneumoperioneum with CO2 and Trendelenburg position, which may have adverse cardiopulmonary effects. A new ventilation mode; pressure-controlled ventilation with volume guaranteed mode (PCV-VG) delivers constant tidal volume with constant inspiratory pressure, using a decelerating flow pattern. This prospective, randomized study is designed to compare the effects of PCV-VG, volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV) on respiratory and hemodynamic variables in patients undergoing Robot-assisted hysterectomy.

DETAILED DESCRIPTION:
1. Total 60 patients with American Society of Anesthesiologists physical status I-II who underwent Robot-assisted hysterectomy were enrolled.
2. All patients were fasted for 8 hours before the surgery and were premedicated with intramuscular glycopyrrolate 0.2 mg. Anesthesia was induced with intravenous remifentanil (0.1-0.2 ug/kg/min), propofol (1.5-2 mg/kg) and rocuronium (0.6 mg/kg) and maintained with sevoflurane (2.0-2.5 vol%) in inspired oxygen fraction with 0.5, remifentanil (0.05-0.3 ug/kg/min) and vecuronium (0.03-0.05 mg/kg/hr).
3. A 20 G catheter was inserted into the radial artery to monitor continuous arterial pressure and hemodynamic variables (cardiac output, cardiac index, stroke volume, stroke volume index, and stroke volume variation) monitoring.
4. All patients were ventilated with a Datex-Ohmeda Ventilator (S/5 AVANCE). Patients were randomized to receive VCV (n=20), PCV (n=20), or PCV-VG (n=20) mode. The tidal volume was set to deliver 8 mL/kg of ideal body weight. The respiratory rate(RR) was adjust to maintain end tidal CO2 (ETCO2) 32-37 mmHg.
5. Hemodynamic variables (mean blood pressure, heart rate, cardiac output, cardiac index, stroke volume, stroke volume index, and stroke volume variation) , respiratory variables (saturation, RR, ETCO2, peak airway pressure, mean airway pressure and lung dynamic compliance) and arterial gas analyses were recorded at 4 stages: (1) 15 minutes after induction in supine position, (2) 30 minutes after pneumoperitoneum and Trendelenburg position, (3) 60 minutes after pneumoperitoneum and Trendelenburg position, (4) 15 minutes after pneumoperitoneum withdrawal in supine position.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for Robot-assisted hysterectomy
* American Society of Anesthesiologists physical status I-II

Exclusion Criteria:

* Age under 20 years old or over 65 years old
* Body mass index > 30 kg/m2
* Systolic blood pressure < 100 mmHg
* Heart rate < 60 bpm
* Uncompensated cardiac disease
* FEV1 < 60%
* Hypoxemia (PaO2 < 60 mmHg or oxygen saturation < 90%)

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Peak airway pressure | 2-3 hours through the surgery
  The highest level of pressure applied to the lung during inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Eun Young Park, MD, Study Director — Hallym Univesity Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Dongan-gu, South Korea

REFERENCES:
- [Background] Assad OM, El Sayed AA, Khalil MA. Comparison of volume-controlled ventilation and pressure-controlled ventilation volume guaranteed during laparoscopic surgery in Trendelenburg position. J Clin Anesth. 2016 Nov;34:55-61. doi: 10.1016/j.jclinane.2016.03.053. Epub 2016 May 2. PMID 27687346
- [Background] Dion JM, McKee C, Tobias JD, Sohner P, Herz D, Teich S, Rice J, Barry ND, Michalsky M. Ventilation during laparoscopic-assisted bariatric surgery: volume-controlled, pressure-controlled or volume-guaranteed pressure-regulated modes. Int J Clin Exp Med. 2014 Aug 15;7(8):2242-7. eCollection 2014. PMID 25232415
- [Background] Pu J, Liu Z, Yang L, Wang Y, Jiang J. Applications of pressure control ventilation volume guaranteed during one-lung ventilation in thoracic surgery. Int J Clin Exp Med. 2014 Apr 15;7(4):1094-8. eCollection 2014. PMID 24955188
- [Background] Ogurlu M, Kucuk M, Bilgin F, Sizlan A, Yanarates O, Eksert S, Karasahin E, Cosar A. Pressure-controlled vs volume-controlled ventilation during laparoscopic gynecologic surgery. J Minim Invasive Gynecol. 2010 May-Jun;17(3):295-300. doi: 10.1016/j.jmig.2009.10.007. Epub 2010 Mar 19. PMID 20303833
- [Background] Kim MS, Soh S, Kim SY, Song MS, Park JH. Comparisons of Pressure-controlled Ventilation with Volume Guarantee and Volume-controlled 1:1 Equal Ratio Ventilation on Oxygenation and Respiratory Mechanics during Robot-assisted Laparoscopic Radical Prostatectomy: a Randomized-controlled Trial. Int J Med Sci. 2018 Oct 20;15(13):1522-1529. doi: 10.7150/ijms.28442. eCollection 2018. PMID 30443174